CLINICAL TRIAL: NCT02332174
Title: Pharmacokinetics and Tolerability of Rufinamide Following Single and Multiple Oral Doses and Effect of Food on Pharmacokinetics in Healthy Chinese Subjects
Brief Title: Pharmacokinetics and Tolerability of Rufinamide in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Weiyong Li, Institute of Clinical Pharmacy, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TJXH-Rufi
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Seizures
Keywords: pharmacokinetics; food effect; sex effect; tolerability
MeSH Terms: conditions — Seizures | interventions — rufinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 200-mg group (Experimental): Ten healthy subjects were administered a single oral dose of 200 mg rufinamide tablets in fasted and fed state at day 1 and then received repeated oral doses of rufinamide (200 mg) once daily for 6 days.
  Interventions: Drug: rufinamide
- 400-mg group (Experimental): Ten healthy subjects were administered a single oral dose of 400 mg rufinamide tablets in fasted state.
  Interventions: Drug: rufinamide
- 800-mg group (Experimental): Ten healthy subjects were administered a single oral dose of 800 mg rufinamide tablets in fasted state.
  Interventions: Drug: rufinamide
- 1200-mg group (Experimental): Ten healthy subjects were administered a single oral dose of 1200 mg rufinamide tablets in fasted state.
  Interventions: Drug: rufinamide

INTERVENTIONS:
Drug: rufinamide — comparison of different doses, sex and medication conditions
  Other Names: 106308-44-5

SUMMARY:
The purpose of this study was to determine the pharmacokinetic (PK) and safety profile of single and multiple doses of rufinamide. The effects of food and sex on the PK properties of rufinamide in these Chinese volunteers were also evaluated.

DETAILED DESCRIPTION:
This single- and multiple-dose, randomized, open-label study was conducted in healthy Chinese subjects. In the single-dose study, volunteers were randomly assigned to 4 dose groups and received a single dose of 200, 400, 800, 1200 mg rufinamide tablets under fasted condition. An additional food effect study was performed in the 200-mg dose group by assessing changes in PK parameters after high-fat diet. In the multiple-dose study, 10 subjects were administered 200-mg rufinamide formulation twice daily for 6 consecutive days. LC-MS/MS method was applied to determine plasma concentration of rufinamide. Tolerability was assessed based on investigator inquiries, spontaneous reports, and clinical evaluations such as standard laboratory tests, vital signs, physical examinations and 12-lead electrocardiography.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between19 and 24 kg/m2
* negative for HIV and hepatitis B
* had no clinicallyimportant findings on health tests
* thorax radiography and ECG with no abnormalities
* normal blood pressure values
* heart rate

Exclusion Criteria:

* any drug treatment within 2 weeks before starting the study
* participation in another clinical study within the previous 3 months
* alcoholism and smoking
* pregnancy
* breast-feeding
* hypocalcemia
* blood donation or participation in other clinical trials within 3 months before enrollment in the study
* sitting blood pressure <80/50 mm Hg or >140/100 mm Hg
* A ventricular rate <60 beats/min or >100 beats/min at rest

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC | three days
  the area under the concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, PhD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology